CLINICAL TRIAL: NCT03748407
Title: Determination of Baseline Thyroid Status Values
Brief Title: Determination of Baseline Thyroid Status Values in French Adult Population
Acronym: THYRBECK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-040
Record Dates: First submitted 2018-10-30; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dosages in Healthy volunteers (Other): Only one arm : healthy volunteer blood donors. Performing a blood test for the determination of parameters that explore thyroid status : only once.
  Absence of other healthy volunteers group all healthy volunteers have a blood test performed in the same way.
  Interventions: Other: Dosages of Thyroid parameters

INTERVENTIONS:
Other: Dosages of Thyroid parameters — Dosages of the following parameters: TSH, FT4 FT3, TGAb (Tyroglobulin antibody) , TPO Ab (ThyroPeroxydase Antibody)

SUMMARY:
The objective of this study is to establish reference values in the general population from a Beckman Coulter DxI chemiluminescence assay.

Indeed, the lack of harmonization of the methods of the dosage remains a major difficulty to optimize the management of patients with thyroid disease.

This supplier has recently optimized its dosing kit according to the 3rd international standard of the WHO (IRB 81/565) for the TSH (Thyroid Stimulating Hormon).

It is necessary to carry out a study of the distribution of the values of this TSH within our metropolitan population. The current data proposed by the supplier come from a study of a North American population.

investigators propose to define usual values for thyroid status markers (TSH, FT4 [free thyroxine], FT3 [free triiodothyroxine]) from healthy EFS (French Blood Establishment) donors who meet the standard exclusion criteria for this type of study.

ELIGIBILITY:
Inclusion Criteria:

* Donors (18-70 years old) volunteers at EFS

Exclusion Criteria:

* pregnancy,
* known antecedents of thyroid diseases (goiter, nodule, hypo or hyperthyroidism),
* current antithyroid treatment (neomercazole [Thyrozol(r)], levothyroxyn LT4 [levothyrox(r)], ...),
* cardiac treatment with amiodarone (cordarone(r)),
* injection of iodinated contrast medium less than 1 month old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-11-30 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the usual values of TSH | baseline
  Determination of the usual values of TSH after assays on DxI automaton of the Beckman Company according to the standardization 3rd international standard (IRB 81/565)
Determination of the usual values of FT4 | baseline
  Determination of the usual values of FT4 after assays on DxI automaton of the Beckman Company according to the standardization 3rd international standard (IRB 81/565)
Determination of the usual values of FT3 | baseline
  Determination of the usual values of FT3 after assays on DxI automaton of the Beckman Company according to the standardization 3rd international standard (IRB 81/565)